CLINICAL TRIAL: NCT02348931
Title: Investigation of the Effect of a Customized Nasal Brace on Nasal Deformities With or Without Prior Surgery
Brief Title: Clinical Effect of a Nasal Former in Nasal Deformities
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT_12_05_2013; 2013-0021 (Other: Ethics Commission of Zurich)
Record Dates: First submitted 2014-03-21; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Nose Deformity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Surgery plus device (Nasella) (Active Comparator): Person in need of surgery has cast for one week, then use of customized nasal brace for nose (Nasella) deformities during 8 weeks.
  Interventions: Device: Use of customized nasal brace (Nasella) for nose deformities; Procedure: corrective surgery
- Surgery, no device thereafter (Experimental): Person in need of surgery has cast for 1 week; thereafter no use of customized nasal brace (Nasella) .
  Interventions: Procedure: corrective surgery
- Only device (Nasella) (Active Comparator): No need for surgery; use of customized nasal brace (Nasella) for nose deformities is made to improve look (cosmetic reason).
  Interventions: Device: Use of customized nasal brace (Nasella) for nose deformities

INTERVENTIONS:
Device: Use of customized nasal brace (Nasella) for nose deformities
  Arms: Only device (Nasella); Surgery plus device (Nasella)
Procedure: corrective surgery
  Arms: Surgery plus device (Nasella); Surgery, no device thereafter

SUMMARY:
Investigation of the effect of customized nasal braces in the correction of nasal deformities with and without prior corrective surgery.

* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria:

* Healthy adults with skewed, humped or broad nose, who are able to attend all follow-ups

Exclusion criteria:

* Inability to keep the research plan
* Allergies to components of the nasal brace
* Diseases of the bone metabolism
* Medication affecting bone metabolism
* Drugs or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Skewed nose: Deviation from the 0° axis in the coronar plain (Philtrum-Glabella line). | 9 Weeks after surgery
  The deviation from a perfect line (0 axis) is measured and compared to control group
Humped nose: Deviation from the 0° axis in the sagittal plain (line from nose root to tip). | 9 Weeks after surgery
  The deviation from a perfect line (0 axis) is measured and compared to control group
Broad nose: Appealing proportion of nose width to eye-corner distance. | 9 weeks after surgery
  The deviation from a perfect line (0 axis) is measured and compared to control group
Skewed nose: Deviation from the 0° axis in the coronar plain (Philtrum-Glabella line). | 14 months of treatment with Nasella
  The improvement in degrees compared to study start
Humped nose: Deviation from the 0° axis in the sagittal plain (line from nose root to tip). | 14 months of treatment with Nasella
  The improvement in degrees compared to study start
Broad nose: Appealing proportion of nose width to eye-corner distance. | 14 months of treatment with Nasella
  The improvement of proportion of width compare to study start

SECONDARY OUTCOMES:
Subjective Satisfaction | 9 weeks postoperatively
Subjective Satisfaction | 14 months of treatment
Doctors assessment of various appearances | 9 weeks postoperatively
Doctors assessment of various appearances | 14 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Roth, Dr. med., Principal Investigator — University Hospital Zurich, Department of Otorhinolaryngology
Locations (1):
- University Hospital Zurich, Department of Otorhinolaryngology, Zurich, Canton of Zurich, Switzerland